CLINICAL TRIAL: NCT04774991
Title: Azithromycin for Child Survival in Niger: Delivery Trial
Acronym: AVENIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Programme National de Santé Oculaire, Ministère de la Santé Publique du Niger (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-28387B
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Mortality; Child Health; Implementation
MeSH Terms: interventions — Azithromycin; Suspensions

STUDY DESIGN:
Intervention Model Description: The AVENIR delivery trial is a two-armed, cluster-randomized trial in the Dosso region in Niger. 80 Communities will be randomized in a 1:1 allocation to either door-to-door delivery or fixed-point delivery of azithromycin to children 1-59 months of age.
Masking Description: In the delivery trial, participants, implementers, and outcome assessors will not be actively masked from the delivery approach given the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithro 1-59 fixed point (Active Comparator): Azithromycin distribution to children 1-59 months of age using a fixed-point delivery approach via existing community health workers
  Interventions: Drug: Azithromycin for Oral Suspension
- Azithro 1-59 door-to-door (Active Comparator): Azithromycin distribution to children 1-59 months of age using a door-to-door delivery approach via existing community health workers
  Interventions: Drug: Azithromycin for Oral Suspension

INTERVENTIONS:
Drug: Azithromycin for Oral Suspension — Azithromycin will be administered as a single dose in oral suspension form for children as follows:
  * Single-dose of 20mg/kg in children (up to the maximum adult dose of 1g)
  * For children 1 to <12 months of age, weight-based dosing will be used
  * For children 12 to 59 months of age, height-based dosing will be used via height-stick approximation as currently performed by Niger's trachoma program.
  Other Names: Zithromax

SUMMARY:
This cluster-randomized trial aims to compare the impact of different delivery approaches to azithromycin distribution on coverage, costs, and feasibility outcomes. The investigators hypothesize that door-to-door delivery will have higher coverage and costs and similar feasibility and acceptability compared to fixed-point delivery.

DETAILED DESCRIPTION:
Azithromycin distribution has been shown to reduce mortality in children 1-59 months. This trial aims to contribute evidence on viable approaches to implementation as high mortality countries consider this intervention to improve child survival. From a pool of eligible rural and peri-urban communities in the Dosso Region in Niger, 80 will be randomly selected and randomized to receive door-to-door or fixed-point delivery of a single dose of azithromycin distribution to children 1-59 months of age via community health workers biannually. Treatment coverage, costs and cost-effectiveness, and feasibility and acceptability will be compared by arm.

ELIGIBILITY:
Inclusion Criteria:

At the community-level, eligibility includes:

* Location in one of the 80 Dosso communities randomly selected for the delivery trial
* Population 250 to 2,499*
* Distance > 5 km from the district headquarters town
* Verbal consent of community leader(s)

At the individual-level, eligibility includes:

* Age 1-59 months
* Primary residence in a study community
* Verbal consent of caregiver/guardian for study participation
* Weight ≥ 4 kg

Exclusion Criteria:

At the community-level, eligibility includes:

* Inaccessible or unsafe for study team
* "Quartier" designation on national census *Population size as estimated from the most recent national census or projections

At the individual-level, eligibility includes:

• Known allergy to macrolides

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10925 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Treatment Coverage | 6 months
  Treatment coverage as defined by the number of doses of azithromycin administered in each community divided by the total eligible population

SECONDARY OUTCOMES:
Program Costs | 6 months
  Program costs as captured by routine administrative data collection during the study period and by micro-costing activities
Fidelity of intervention rollout | 6 months
  Fidelity of intervention rollout reported as the percent of protocol steps with complete adherence by the field team
Acceptability of intervention | 6 months
  Participant and provider perception of acceptability of delivery approaches as measured by surveys conducted post-distribution

CONTACTS AND LOCATIONS:
Overall Officials: Tom M Lietman, MD, Principal Investigator — University of California, San Francisco; Kieran S O'Brien, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Program National de Santé Oculaire, Niamey, Niger

IPD SHARING:
Plan to Share IPD: Yes
Data underlying outcomes publications will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data will be made available after publication of the outcomes and will be made available indefinitely
Access Criteria: Once made available, the data will be open access.

REFERENCES:
- [Derived] Arzika AM, Maliki R, Amza A, Karamba A, Gallo N, Aichatou B, Sara II, Beidi D, Haroun LM, Oumarou F, Lebas E, Peterson B, Colby E, Nguyen W, Liu Z, Fitzpatrick MC, Arnold BF, Lietman TM, O'Brien KS; AVENIR Study Group. Comparison of door-to-door and fixed-point delivery of azithromycin distribution for child survival in Niger: A cluster-randomized trial. PLOS Glob Public Health. 2023 Nov 15;3(11):e0002559. doi: 10.1371/journal.pgph.0002559. eCollection 2023. PMID 37967058